CLINICAL TRIAL: NCT01627509
Title: Comparison of Modern Premixed Insulin and Basal-Bolus Regimens on Blood Glucose Control Using CGMS Device in Optimally-controlled Subjects With DM2.
Brief Title: Comparison of Two Insulin Regimens in Optimally-controlled Patients With DM2.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-10-7894-JI-CTIL
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus 2 Type
Keywords: continuous glucose monitoring system; hypoglycemia; insulin regimen; basal bolus therapy; modern premixed insulin; diabetes control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Intensive Insulin Therapy (IIT) may be given in Type 2 Diabetes (T2DM) in two different ways :

* as Basal/bolus therapy (B/B) in four-five injections per day .
* as Modern Premixed Insulins( MPI's) three times per day . The better diabetes control is achieved, the more likely patient would suffer from hypoglycemic episodes. We propose that the probability of hypoglycemia and its severity has no difference in two main insulin therapy schemes mentioned above.

The objective of the study is to compare the incidence of hypoglycemia and its severity in well-controlled ( HBA1C less than 7%) diabetic individuals treated by two different regimens, through analysis of data received by Continuous Glucose Monitoring (CGM, Free Style Navigator).

ELIGIBILITY:
Major Inclusion Criteria:

* Diabetes Mellitus Type 2 diagnosis confirmed by endocrinologist.
* Diabetes Mellitus Type 2 history of one year at least.
* HAb1C < 7% and less
* Age 18-80 yrs
* Normal Liver function tests

Major Exclusion Criteria:

* History of substance use
* Pregnancy or breastfeeding mothers
* Abnormal liver or kidney functional tests
* Type 1 Diabetes or LADA
* any active disease ( like viral) at the period of investigation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 Subjects with 1 year and more of T2DM history , with two consistent HbA1C values of 7% or less - according to the blood tests within last six months.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - The Institute of Endocrinology, Sheba Medical Center, Tel Litwinsky, Gush Dan
  - Sheba Medical Center, Tel Litwinsky